CLINICAL TRIAL: NCT00293475
Title: A Phase I/II Study of Patients With Newly Diagnosed Primary Central Nervous System Lymphoma Treated With Methotrexate/BBBD, and Adding Rituximab (an Anti CD-20 Antibody) and Carboplatin, to the Treatment Regimen
Brief Title: Methotrexate, Mannitol, Rituximab, and Carboplatin in Treating Patients With Newly Diagnosed Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00001012; NCI-2013-00787 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEM-08059-LX (Other: OHSU Knight Cancer Institute); CR00022596 (Other: OHSU IRB); MR00041596 (Other: OHSU IRB); MR00045915 (Other: OHSU IRB Number); SOL-05025-LM (Other: OHSU Knight Cancer Institute); SOL-05025-L (Other: OHSU Knight Cancer Institute); IRB00001012 (Other: OHSU Knight Cancer Institute); R01CA137488 (NIH)
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Central Nervous System Lymphoma
MeSH Terms: interventions — Carboplatin; Mannitol; Methotrexate; merphos; Rituximab; CT-P10; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (rituximab, mannitol, methotrexate, carboplatin) (Experimental): Patients receive rituximab IV over 5 hours on day 1, mannitol IA, methotrexate IA over 10 minutes, and carboplatin IA over 10 minutes on days 2 and 3. Patients then receive sodium thiosulfate IV over 15 minutes at 4 and 8 hours after carboplatin. Treatment repeats monthly for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Mannitol; Drug: Methotrexate; Other: Quality-of-Life Assessment; Biological: Rituximab; Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Carboplatin — Given IA
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Mannitol — Given IA
  Other Names: D-Mannitol; Mannitol, D-; Osmitrol; Resectisol
Drug: Methotrexate — Given IA
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Sodium Thiosulfate — Given IV
  Other Names: Cyanide Antidote Package; Disodium Thiosulfate; S-Hydril; Sodium Hyposulfate; Sodium Thiosulfate Pentahydrate; Sodium Thiosulphate; Sodothiol; Thiosulfate, Sodium, Pentahydrate; Thiosulfuric Acid Disodium Salt

SUMMARY:
This phase I/II trial studies the side effects of methotrexate, mannitol, rituximab, and carboplatin and to see how well they work in treating patients with primary central nervous system lymphoma. Drugs used in chemotherapy, such as methotrexate and carboplatin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Osmotic blood-brain barrier disruption uses mannitol to open the blood vessels around the brain and allow cancer-killing substances to be carried directly to the brain. Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Giving methotrexate, mannitol, rituximab, and carboplatin together may be an effective treatment for primary central nervous system lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicities of a treatment regimen consisting of rituximab (intravenously [IV]) the day prior to methotrexate (intra-arterially [IA]), and carboplatin (IA) in conjunction with blood-brain barrier disruption (BBBD) and delayed sodium thiosulfate (IV).

II. To demonstrate, adding a monoclonal antibody and carboplatin to methotrexate BBBD, that a 45% rate of complete response (CR) within the first 3 months of treatment is achieved, while excluding a CR rate as low as 30%.

SECONDARY OBJECTIVE:

I. To estimate the response rate (counting all CRs), the two-year overall survival and the two-year event-free survival, as baselines for subsequent trials.

OUTLINE:

Patients receive rituximab IV over 5 hours on day 1, mannitol IA, methotrexate IA over 10 minutes, and carboplatin IA over 10 minutes on days 2 and 3. Patients then receive sodium thiosulfate IV over 15 minutes at 4 and 8 hours after carboplatin. Treatment repeats monthly for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 months, then every 2 months for 2 years, every 6 months for 1 year, and then annually for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathologic confirmation of intermediate or high-grade primary central nervous system lymphoma (PCNSL) as documented by brain biopsy, or cytology (analysis from cerebral spinal fluid [CSF] or vitrectomy), and cluster of differentiation 20 (CD20) positive; whenever possible, the tumor should be characterized by immunophenotype
* Subjects must be =< 90 days from diagnosis of PCNSL in the brain or spine; time from pathologic diagnosis to initiation of treatment should be specified; subjects with history of only ocular lymphoma are eligible if < 90 days since documented brain parenchymal disease (by imaging or by biopsy)
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance score =< 3 (Karnofsky >= 30)
* Hematocrit >= 25% (may be reached by transfusion) (performed within 14 days of registration)
* White blood cell count >= 2.5 x 10^3/mm^3 (performed within 14 days of registration)
* Absolute granulocyte count >= 1.2 x 10^3/mm^3 (performed within 14 days of registration)
* Platelets >= 100 x 10^3/mm^3 (or >= lower limit of institutional normal value) (performed within 14 days of registration)
* Calculated creatinine clearance (Cr Cl) >= 50 ml/min (performed within 14 days of registration); eligible for full dose methotrexate
* Calculated Cr Cl >= 30 ml/min (performed within 14 days of registration); eligible for reduced dose methotrexate
* Bilirubin =< 2.0 x upper limit of institutional normal value (performed within 14 days of registration)
* The subject may have had other systemic chemotherapy for PCNSL during the 90 days since PCNSL diagnosis; prior systemic chemotherapy must have been given at least 4 weeks prior to study entry (6 weeks for nitrosourea agents), with the exceptions of methotrexate and rituximab which may have been given at least 10 days prior; ocular lymphoma treatment may have been given any time prior to study entry; if the subject has undergone treatment for parenchymal disease and the parenchymal disease has progressed on a stable or increasing dose of steroids, the subject is not eligible for enrollment
* Sexually active women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study treatment and for the duration of study treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Subjects with a bone marrow biopsy which shows microscopic, low-level involvement of lymphoma are eligible
* Subject with seropositivity for hepatitis B or hepatitis C must be cleared by hepatology service prior to participating in treatment protocol

Exclusion Criteria:

* Prior cranial or spinal radiotherapy
* Subjects with radiographic signs of excessive intra-cranial mass effect with associated rapid neurologic deterioration, and/or spinal block, are unsafe to undergo BBBD chemotherapy and are not eligible
* Uncontrolled (over the last 30 days), clinically significant confounding medical conditions
* Seropositivity for the human immunodeficiency virus
* Systemic lymphoma
* Subjects who have a positive serum human chorionic gonadotropin (hCG), are pregnant or lactating are ineligible
* Known allergy to any of the study agents
* Subjects who are at significant risk for general anesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2005-10-14 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicities, assessed using National Cancer Institute Common Toxicity Criteria for Adverse Events version 3.0 (Phase I) | Within 2 months of completion of study treatment
CR rate (Phase II) | Within the first 3 months of treatment

SECONDARY OUTCOMES:
Overall survival | From entry onto study until death from any cause, assessed at 2 years
  Kaplan-Meier estimates of these survival distributions will be plotted. Descriptive stratifications of these survival distributions by baseline characteristics will be evaluated using the log-rank statistic. If there are multiple predictors of these outcomes, Cox proportional hazard models will be fit to these data to determine which predictors are independent of others in a multi-variable model.
Event-free survival | From entry onto study until death or progression of disease, assessed at 2 years
  Kaplan-Meier estimates of these survival distributions will be plotted. Descriptive stratifications of these survival distributions by baseline characteristics will be evaluated using the log-rank statistic. If there are multiple predictors of these outcomes, Cox proportional hazard models will be fit to these data to determine which predictors are independent of others in a multi-variable model.

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, Principal Investigator — OHSU Knight Cancer Institute
Locations (4):
- United States (4):
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - OHSU Knight Cancer Institute, Portland, Oregon